CLINICAL TRIAL: NCT03842358
Title: Improving Diagnostic US for Reduction of Benign Breast Biopsies Using US-guided Optical Tomography
Brief Title: Diagnostic US for Reduction of Benign Breast Biopsies Using US-guided Optical Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201707042; 1R01CA228047-01A1 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-02-15 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- US-DOT (US/NIR) Imaging (Experimental): * US-DOT (US/NIR) Imaging Exam
  * Breast biopsy or FNA performed (standard of care)
  * A hand-held hybrid probe will be used for the scans
  Interventions: Device: Hand-held hybrid probe

INTERVENTIONS:
Device: Hand-held hybrid probe — Consists of a commercially available US transducer located in the middle and near-infrared source and detector optical fibers distributed at the periphery

SUMMARY:
Ultrasound-guided diffuse optical tomography (DOT) has demonstrated its potential role in differentiating malignant and benign breast abnormalities and in predicting and monitoring the neoadjuvant chemotherapy (NAC) response of breast cancer. This unique approach employs a commercial ultrasound (US) transducer and near infrared (NIR) optical imaging sensors mounted on a hand-held US probe. The co-registered US is used for lesion localization, and optical sensors are used for imaging tumor related vascularity.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ≥ 18 years old with ultrasound visible breast abnormalities (BI-RADS 3*, 4A, 4B, 4C, and 5) referred for ultrasound-guided core needle biopsy or fine needle aspiration

  *note that while a BI-RADS 3 assessment is probably benign, a subset of patients with this assessment choose to undergo biopsy rather than follow up imaging).
* Willing and able to provide informed consent

Exclusion Criteria:

* Lesions located in the darkly pigmented nipple-areolar complex area
* Subjects with breast implants
* Abnormality in the mirror image location of the contralateral breast.
* Additional abnormalities in the same region of the breast that would be included in US-guided DOT imaging of the abnormality undergoing biopsy
* Previous breast irradiation of the mirror image location of the contralateral breast
* Lesions located at previous biopsy sites when biopsy occurred within the last six months.
* Pregnancy
* Superficial abnormalities located entirely within (i.e. less than) 5mm of the overlying skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Bennett, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol states that there are two phases: phase I - training set and phase 2 - prospective trial. For the training set, the readers underwent an approximately 60-minute training session using a tool created from a pre-existing representative DOT findings in patients who had previously undergone US-guided DOT and who had a spectrum of documented benign and malignant pathology. Those patients were not consented or enrolled in this study and are not included in the presented data.
Period: Overall Study
Arm/Group | US-DOT (US/NIR) Imaging
Started | 298
Completed | 286
Not Completed | 12
Not completed — Poor DOT probe contact with breast | 2
Not completed — DOT system problem | 1
Not completed — Switched to x-ray guided biopsy | 3
Not completed — No biopsy after physician review | 4
Not completed — Patient withdrew | 2

BASELINE CHARACTERISTICS:
Population: The protocol states that there are two phases: phase I - training set and phase 2 - prospective trial. For the training set, the readers underwent an approximately 60-minute training session using a tool created from a pre-existing representative DOT findings in patients who had previously undergone US-guided DOT and who had a spectrum of documented benign and malignant pathology. Those patients were not consented or enrolled in this study and are not included in the presented data.
Arm/Group | US-DOT (US/NIR) Imaging
Number analyzed (Participants) | 298
Age, Continuous [Median (Full Range); unit: years] | 50 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 287
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 86
  White | 201
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 298

OUTCOME MEASURES:

1. Primary Outcome: Impact of US-guided DOT on the Potential Reduction of Benign Biopsies as Measured by Comparing the Reads With a Non- Suspicious Assessment of Conventional Imaging (CI) Alone Versus CI & US-DOT
Description: -BI-RADS scores without and then with optical data will be rendered by study radiologists. Radiologists will be blinded to the biopsy exam and pathology outcomes. Optical data including total Hemoglobin concentration will be provided by the bioengineering team. Benign biopsy reduction will be calculated as the proportion of reads (CI & US-DOT subtract CI) with a non- suspicious assessment, i.e. BIRADS 2 'benign' or BIRADS 3 'probably benign', divided by the denominator of total reads with no cancer demonstrated at biopsy. US-guided core biopsy results and subsequent surgical pathology (if present) will be entered by the study pathologist.
Time Frame: Completion of enrollment for all patients (61 months), the imaging session took approximately 1 hour for the participating patient
Measure: Count of Units; unit: BIRADS assessments
Units Other Than Participants: BIRADS assessments
Arm/Group | US-DOT (US/NIR) Imaging
Number analyzed (Participants) | 286
Number analyzed (BIRADS assessments) | 628
BIRADS assessments | 148

2. Primary Outcome: Impact of US-guided DOT as an Adjunct to Conventional Breast Imaging on Maintaining High Sensitivity as Measured by Comparing the False Negative Rate or Missing Malignancy of Conventional Imaging (CI=US +/- Mammography) Alone Versus CI & US-DOT
Description: -BI-RADS scores without and then with optical data will be rendered by study radiologists. Radiologists will be blinded to the biopsy exam and pathology outcomes. Optical data including total Hemoglobin concentration will be provided by the bioengineering team. The engineering team is also blinded to the biopsy exam and pathology outcomes. The False Negative Rate will be calculated as the proportion of reads with a non-suspicious assessment i.e. BIRADS 2 'benign' or BIRADS 3 'probably benign', who have cancer (defined as Invasive cancer or Ductal Carcinoma In Situ) demonstrated at biopsy divided by the denominator of all reads with cancer. US-guided core biopsy results and subsequent surgical pathology (if present) will be entered by the study pathologist.
Time Frame: as for outcome 1
Measure: Count of Units; unit: BIRADS assessments
Units Other Than Participants: BIRADS assessments
Arm/Group | US-DOT (US/NIR) Imaging
Number analyzed (Participants) | 286
Number analyzed (BIRADS assessments) | 329
BIRADS assessments | 5

3. Primary Outcome: Assess the Impact of Adjunctive US-guided DOT Data in the Management of Discordant Pathology Results
Time Frame: as for outcome 1
Population: There were not any cases that were considered discordant in clinical practice as such there was not any data to present for this outcome measure.
Arm/Group | US-DOT (US/NIR) Imaging
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events that occurred within 24 hours of an NIR/US exam were collected. All-cause mortality was collected through 24 hours of the NIR/US exam.
Description: The protocol states that there are two phases: phase I - training set & phase 2 - prospective trial. For the training set, the readers underwent a training session using a tool created from a pre-existing DOT findings in patients who had previously undergone US-guided DOT and who had a spectrum of documented benign and malignant pathology. Those patients were not consented or enrolled in this study and are not included in the data.
  Non-serious adverse events were not collected for the patients.
Arm/Group | US-DOT (US/NIR) Imaging
All-Cause Mortality (participants affected / at risk) | 0/286
Serious Adverse Events (participants affected / at risk) | 0/286
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03842358/Prot_SAP_001.pdf
  • Informed Consent Form (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT03842358/ICF_000.pdf